CLINICAL TRIAL: NCT06801834
Title: A Global, Multicenter, Randomized, Open-label, Phase 3 Study of Sacituzumab Govitecan Versus Standard of Care (SOC) in Participants With Previously Treated Extensive Stage Small Cell Lung Cancer (ES-SCLC)
Brief Title: Study of Sacituzumab Govitecan Versus Standard of Care in Participants With Previously Treated Extensive Stage Small Cell Lung Cancer
Acronym: EVOKE-SCLC-04
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-600-6165; 2024-515884-69 (Other: European Medicines Agency)
Record Dates: First submitted 2025-01-24; First posted 2025-01-30 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Extensive Stage Small Cell Lung Cancer (ES-SCLC)
MeSH Terms: interventions — sacituzumab govitecan; Topotecan; amrubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Group A: SG (Experimental): Participants assigned to treatment group A will receive SG 10 mg/kg intravenous (IV) infusion on Days 1 and 8 of a 21-day cycle. Participants will receive study drug until progressive disease (PD), death, unacceptable toxicity, or another treatment discontinuation criterion is met.
  Interventions: Drug: Sacituzumab Govitecan (SG)
- Treatment Group B: Topotecan or Amrubicin (Japan only) (Experimental): Participants assigned to treatment group B will receive Topotecan 1.5 mg/m^2 daily on Days 1 to 5 of a 21-day cycle.
  Japan participants assigned to treatment group B will have the option to receive Topotecan 1.5 mg/m^2 daily on Days 1 to 5 of a 21-day cycle, or Amrubicin 40 mg/m^2 daily on Days 1 to 3 of a 21-day cycle.
  Participants will receive study drug until PD, death, unacceptable toxicity, or another treatment discontinuation criterion is met.
  Interventions: Drug: Topotecan; Drug: Amrubicin (Japan only)

INTERVENTIONS:
Drug: Sacituzumab Govitecan (SG) — Administered intravenously
  Other Names: Trodelvy®; GS-0132; IMMU 132
  Arms: Treatment Group A: SG
Drug: Topotecan — Administered intravenously
  Arms: Treatment Group B: Topotecan or Amrubicin (Japan only)
Drug: Amrubicin (Japan only) — Administered intravenously
  Arms: Treatment Group B: Topotecan or Amrubicin (Japan only)

SUMMARY:
The goal of this clinical study is to learn more about the study drug sacituzumab govitecan (SG; Trodelvy®; GS-0132; IMMU 132), versus standard of care (SOC) in participants with previously treated extensive stage small cell lung cancer (ES-SCLC).

The primary objectives of this study are to compare the effect of SG to SOC on objective response rate (ORR) as assessed by blinded independent central review (BICR) according to the Response Evaluation Criteria in Solid Tumors and to compare the effect of SG to SOC on overall survival (OS).

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically confirmed diagnosis of SCLC.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.
* Measurable disease by computed tomography (CT) or magnetic resonance imaging (MRI) as assessed by investigator per RECIST v1.1 criteria.
* Documentation of radiological disease progression after 1 prior line of platinum-containing chemotherapy (defined as at least 2 cycles of treatment) with or without therapy directed against programmed cell death protein 1 (PD-1) or programmed cell death ligand 1 (PD-L1; PD-1 and PD-L1 are hereafter referred to as PD-(L)1) for ES-SCLC.

Key Exclusion Criteria:

* Chemotherapy-free interval (CTFI) time from the last dose of first-line platinum-containing chemotherapy to the occurrence of progressive disease) < 30 days (independent of the immunotherapy maintenance).
* Received any prior treatment with irinotecan, topotecan, SG, SN-38, exatecan derivatives, and similar agents targeting topoisomerase I.
* Untreated central nervous system (CNS) metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they have stable CNS disease (ie, without evidence of progression) for at least 4 weeks prior to enrollment and all neurologic symptoms have returned to baseline, have no evidence of new or enlarging brain metastases, and are taking ≤ 10 mg/day of prednisone or its equivalent.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 695 (Estimated)
Dates: Start 2025-04-04 (Actual); Primary Completion 2029-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to 4.5 years
  ORR is defined as the percentage of participants who have achieved a complete response (CR) or partial response (PR) as assessed by BICR according to RECIST v1.1
Overall Survival (OS) | Up to 4.5 years
  OS is defined as length of time from randomization until the date of death from any cause.

SECONDARY OUTCOMES:
Progression-free Survival (PFS) | Up to 4.5 years
  PFS is defined as the time from date of randomization until disease progression as assessed by BICR according to RECIST v1.1 or death from any cause, whichever comes first.
Duration of Response (DOR) | Up to 4.5 years
  DOR is defined as is measured from the time of first response (CR or PR) as assessed by BICR according to RECIST v1.1, until the date of first documented disease progression or death, whichever comes first
Time to First Deterioration in Shortness of Breath Domain | Up to 4.5 years
  Time to first deterioration is defined as the time from the date of randomization to the first time a participant experienced change from baseline equal to or greater than the prespecified threshold value for deterioration or death.
Time to First Deterioration in Physical Functioning Domain | Up to 4.5 years
  Time to first deterioration is defined as the time from the date of randomization to the first time a participant experienced change from baseline equal to or greater than the prespecified threshold value for deterioration or death.
Percentage of Participants Experiencing Treatment-emergent Adverse Events (TEAEs) | First dose date up to 4.5 years
  TEAE is defined as any AEs occurred during the treatment-emergent period. The treatment-emergent period is defined as the time period from the first dose of study treatment to the earlier of 30 days following the last dose of study treatment or the initiation of subsequent anticancer therapy.
Percentage of Participants Experiencing Clinical Laboratory abnormalities | First dose date up to 4.5 years
  Laboratory abnormality is defined as any value that increases at least 1 toxicity grade from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (196):
- United States (17):
  - Los Angeles Cancer Network, Anaheim, California
  - Hope and Healing Cancer Services, Hinsdale, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Parkview Research Center, Fort Wayne, Indiana
  - IU Health Ball Memorial Hospital and Physicians - Cancer Center - Muncie, Muncie, Indiana
  - Northwest Cancer Centers, Dyer, Kentucky
  - St. Claire Regional Medical Ce, Morehead, Kentucky
  - New Mexico Oncology Hematology Consultants, Ltd, Albuquerque, New Mexico
  - University Hospitals Seidman Cancer Center, Sandusky, Ohio
  - Taylor Cancer Research Foundation, Toledo, Ohio
  - Spoknwrd Clinical Trials Inc., Easton, Pennsylvania
  - Hendrick Health System, Abilene, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Texas Oncology - San Antonio, New Braunfels, Texas
  - The University of Texas Health Science Center at Tyler, Tyler, Texas
  - Gundersen Health System, West Salem, Wisconsin
- Argentina (6):
  - Hospital Britanico de Buenos Aires, Buenos Aires
  - Universidad de Buenos Aires - Facultad de Medicina - Instituto Alexander Fleming (Buenos Aires), Buenos Aires
  - Clinica Colon S.A.A (Clinica y Maternidad Colon) Investigaciones Clinicas de Mar del Plata, Buenos Aires
  - Centro Oncologico de Excelencia (San Juan), San Juan
  - Centro Médico San Roque, San Miguel de Tucumán
  - Sanatorio Parque SA, Santa Fe
- Australia (6):
  - Cancer Care Wollongong, New South Wales, New South Wales
  - Metro North HHS (The Prince Charles Hospital), Queensland, Queensland
  - Gold Coast University Hospital, Southport, Queensland
  - Cancer Research SA, Adelaide, South Australia
  - St Vincent's Hospital Melbourne, Fitzroy, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
- Belgium (4):
  - Grand Hopital de Charleroi, Charleroi
  - Jessa Ziekenhuis, Hasselt
  - AZ Delta, Roeselare
  - Vitaz, Sint-Niklaas
- Brazil (12):
  - Instituto do Cancer do Ceara, Fortaleza Ceara
  - Hospital de Caridade de Ijui, Ijuí
  - Liga Norte-Rio-Grandense Contra o Cancer - Pesquisa Clinica, Natal
  - Hospital Mae de Deus, Porto Alegre
  - Hospital Sao Lucas da PUC Rio Grande do Sul, Porto Alegre
  - IMIP - Instituto de Medicina Integral Professor Fernando Figueira, Recife Pernambuco
  - Grupo Oncoclínicas, Santa Lúcia
  - Centro de Estudos e Pesquisa de Hematologia e Oncologia, Santo André
  - Instituto Hemomed Oncologia e Hematologia, São Paulo
  - Fundação Pio XII - Hospital de Amor, São Paulo
  - HB Onco, São Paulo
  - Hospital Amaral Carvalho, São Paulo
- Canada (5):
  - Royal Victoria Regional Health Centre, Barrie
  - Hamilton Health Sciences - Juravinski Cancer Centre, Hamilton
  - McGill University, Montreal
  - CISSS BSL / Hopital regional de Rimouski, Rimouski
  - Sunnybrook Health Sciences Centre, Toronto
- China (31):
  - Beijing Cancer Hospital, Beijing
  - Jilin Cancer Hospital, Changchun
  - Sichuan Cancer Hospital, Chengdu
  - Chongqing University Cancer Hospital, Chongqing
  - Fujian Medical University Union Hospital, Fuzhou
  - Sun Yat-sen University Cancer Center, Guangzhou
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - The Second Affiliated Hospital of Nanchang University, Jiangxi
  - Affiliated Cancer Hospital of Shandong First Medical University, Jinan
  - The Second Affiliated Hospital of Kunming Medical University, Kunming
  - Linyi Cancer Hospital, Linyi
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - Jiangsu Cancer Hospital, Nanjing
  - Shanghai Chest Hospital, Shanghai
  - Fudan University Shanghai Cancer Center, Shanghai
  - Shanxi Provincial Cancer Hospital, Shanxi
  - Cancer Hospital Chinese Academy of Medical Sciences, Shenzhen Center, Shenzhen
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin
  - Weifang No.2 People's Hospital, Weifang
  - Tongji Hospital, Tongji Medical College of Huazhong University of Science and Technology, Wuhan
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - The First Affiliated Hospital of Xiamen University, Xiamen
  - The First Affiliated Hospital of Xinxiang Medical University, Xinxiang
  - Northern Jiangsu People's Hospital, Yangzhou
  - Henan Provincial Cancer Hospital, Zhengzhou
- France (11):
  - CHU Angers - Hôpital Larrey, Angers
  - Centre Hospitalier Intercommunal de Créteil, Créteil
  - CHU Grenoble Alpes - Hopital Albert Michallon, La Tronche
  - Hôpital Lyon Sud - Hospices Civils de Lyon, Lyon
  - Assistance Publique - Hopitaux de Marseille, Hopital Nord, Marseille
  - Hopital Tenon - Assistance Publique Hopitaux de Paris, Paris
  - Institut Curie, Paris
  - Hopital Haut-Leveque, Pessac
  - CHU Rennes - Hopital Pontchaillou, Rennes
  - Centre Hospitalier Universitaire de Nantes, Saint-Herblain
  - Hopital Saint Joseph - Paris, Saint-Mandé
- Germany (5):
  - Klinikum Chemnitz gGmbH, Chemnitz
  - Klinikum Esslingen GmbH, Klinik fur Kardiologie, Angiologie and Pneumologie, Esslingen am Neckar
  - UKE Hamburg-Eppendorf fur Onkologie, Hamburg
  - Katholisches Marienkrankenhaus gGmbH, Hamburg
  - Johannes Wesling Klinikum Minden, Minden
- Greece (7):
  - Anticancer-Oncology Hospital of Athens 'Agios Sawas' 1st Pathology-Oncology Department, Athens
  - Henry Dunant Hospital Center, 4th Oncology Clinic, Athens
  - Metropolitan Hospital, Athens
  - University General Hospital of Larissa Department of Medical Oncology, Larissa
  - University General Hospital of Patras, Division of Oncology, Rio
  - St Luke's Hospital Oncology Department, Panorama, Thessaloniki
  - Interbalkan Hospital of Thessaloniki, Thessaloniki
- Israel (5):
  - Soroka Medical Center, Beersheba
  - Rambam Health Care Campus, Haifa
  - Hadassah Medical Center, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Galilee Medical Center, Naharyia
- Italy (9):
  - Fondazione IRCCS - Istituto Nazionale dei Tumori di Milano, Aviano
  - IRCCS Candiolo - Istituto di Ricerca, Candiolo
  - Ospedale San Luca - Lucca, Lucca
  - ASST - Grande Ospedale Metropolitano Niguarda, Milan
  - Istituto Nazionale Tumori IRCCS Fondazione G. Pascale Naples, Naples
  - Istituto Nazionale Tumori IRCCS Fondazione G. Pascale, Naples
  - Casa di cura Pederzoli, Peschiera del Garda
  - Istituti di Ricovero e Cura A Carattere Scientifico - Istituti Fisioterapici Ospitalieri, Roma
  - Universita Cattolica del Sacro Cuore, Roma
- Japan (19):
  - Nagoya University Hospital, Aichi
  - Shikoku Cancer Center, Ehime
  - Kyushu University Hospital, Fukuoka
  - Kurume University Hospital, Fukuoka
  - Hiroshima City Hiroshima Citizens Hospital, Hiroshima
  - Hyogo Cancer Center, Hyōgo
  - Kanagawa Cancer Center, Kanagawa
  - Kobe City Medical Center General Hospital, Kobe
  - Sendai Kousei Hospital, Miyagi
  - Niigata University Medical & Dental Hospital, Nigata-shi
  - Okayama University Hospital, Okayama
  - Osaka City General Hospital, Osaka
  - Kansai Medical University Hospital, Osaka
  - Kindai University Hospital, Osaka
  - National Hospital Organization Kinki Chuo Chest Medical Center, Osaka
  - Saitama Prefectural Cancer Center, Saitama
  - Juntendo University School of Medicine Juntendo Clinic, Tokyo
  - Nippon Medical School (all Hospitals), Tokyo
  - The Cancer Institute Hospital of JFCR, Tokyo
- Malaysia (5):
  - Pantai Hospital Kuala Lumpur, Kuala Lumpur
  - Beacon Hospital, Kuala Selangor
  - Sunway Medical Centre, Kuala Selangor
  - Sarawak General Hospital, Kuching
  - University Malaya Medical Centre, Lembah Pantai
- Netherlands (5):
  - Amsterdam UMC, Locatie VUMC, Amsterdam
  - Zuyderland Medisch Centrum, Heerlen
  - Frisius MC location Leeuwarden, Leeuwarden
  - Maastricht University Medical Center, Maastricht
  - Sint Antonius Ziekenhuis, Utrecht
- Norway (2):
  - Haukeland University hospital, Bergen
  - Oslo University Hospital, Oslo
- Poland (5):
  - Uniwersytet Medyczny w Lodzi, Lodz
  - Poznan University of Medical Sciences, Poznan
  - Podkarpackie Centrum Onkologii Rzeszow, Rzeszów
  - Mazowiecki Szpital Wojewódzki im. św. Jana Pawła II w Siedlcach, Siedlce
  - Wojewodzki Szpital Specjalistyczny im. Janusza Korczaka w Słupsku, Stupsk
- Romania (6):
  - Spitalul Clinic Coltea, Bucharest
  - S.C Radiotherapy Center Cluj S.R.L, Cluj-Napoca
  - S.C Centrul de Oncologie S.F Nectarie SRL, Craiova
  - S.C Ovidius Clinical Hospital S.R.L, Ovidiu
  - Spitalul Municipal Ploiesti, Ploieşti
  - S.C Oncomed S.R.L, Timișoara
- South Korea (12):
  - Samsung Changwon Hospital, Changwon-Si
  - Chonnam National University Hwasun Hospital, Gwangju
  - Korea University Anam Hospital, Seongbuk-Gu
  - Seoul National University Bundang Hospital, Seongnam
  - Kangbuk Samsung Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - Yonsei University Severance Hospital, Seoul
  - Gyeongsang National University Hospital, Seoul
  - The Catholic University of Korea, St. Vincent's Hospital, Suwon
  - Ulsan University Hospital, Ulsan
- Spain (15):
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - Hospital Universitari Vall d'Hebron, Barcelona
  - CEIC - Hospital Clinic i Provincial de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - ICO(Instituto Catalan de Oncologia) Badalona - Germans Trias i Pujol, Barcelona
  - Institut Catala d'Oncologia Girona, Girona
  - Complejo Hospitalario de Jaén, Jaén
  - Complejo Hospitalario Universitario Insular Materno-Infantil, Las Palmas de Gran Canaria
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Facultad de Medicina. Universidad Complutense de Madrid, Madrid
  - Hospital Quironsalud Malaga, Málaga
  - Hospital Universitario Virgen de Valme Sevilla, Seville
  - Hospital Universitario Virgen de Valme, Seville
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Universitari i Politecnic La Fe, Valencia
- Taiwan (8):
  - Changhua Christian Hospital, Changhua
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Taipei Veterans General Hospital, Taipei
  - National Taiwan University Cancer Center, Taipei
  - Koo Foundation Sun Yat-Sen Cancer Center, Taipei
  - Chang Gung Memorial Hospital, Linkou, Taoyuan
- The Christie NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study?nctid=NCT06801834